CLINICAL TRIAL: NCT06637189
Title: Protocol with Progestin-primed Ovarian Stimulation (PPOS) from the Beginning of Stimulation Versus Protocol with GnRH Antagonists for Ovarian Stimulation in Patients Undergoing DUOSTIM with Embryo Accumulation for PGT-A.
Acronym: PPDUO
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ginefiv (Other)
Collaborators: Theramex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2306-GFMAD-129-CB; 2023-508769-33 (EudraCT Number)
Record Dates: First submitted 2024-04-25; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Stimulation in the Ovary; Embryo; Oocyte; Oocyte Retrieval; Fertilization in Vitro; Blastocyst; PGT-A
Keywords: duostim; ovarian stimulation; progesterone; GnRH antagonists; PGT-A
MeSH Terms: interventions — ganirelix; Medroxyprogesterone Acetate

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized non-inferiority study. There will be two groups of patients:
  Patients in Group A (PPOS protocol - study group) will start controlled ovarian stimulation with the administration of FSHr gonadotropin at doses between 225 IU-300 IU/day (depending on patient characteristics) + 10 mg medroxyprogesterone/day (IMP).
  Patients in Group B (Short protocol with GnRH antagonists - control group) will start controlled ovarian stimulation with the administration of FSHr gonadotropin at doses between 225 IU-300 IU/day (depending on patient characteristics) and will add treatment with a GnRH antagonist at a dose of 0.25 mg/day from the 6th day of stimulation or when a follicle with a size equal to or greater than 14 mm is present.
  Once the two stimulations typical of the DuoStim strategy are completed, the results obtained in both groups will be compared.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PPOS - study group (Experimental): Patients belonging to this arm will initiate controlled ovarian stimulation by administering FSHr gonadotropin at doses between 225 IU-300 IU/day (according to patient characteristics) + 10mg medroxyprogesterone/day (IMP) from day 2-3 of their menstrual cycle.
  Both groups will continue with the usual regimen of administration of all medications related to Ovarian Stimulation
  Interventions: Drug: Medroxyprogesterone Acetate 10 MG
- GnRH antagonists - control group (Active Comparator): Patients belonging to this arm will initiate controlled ovarian stimulation by administering FSHr gonadotropin at doses between 225 IU-300 IU/day (according to patient characteristics) from day 2-3 of their menstrual cycle, and treatment with the GnRH antagonist at a dose of 0.25 mg/day from the 6th day of stimulation or when a follicle with a size equal to or greater than 14mm is present. Both groups will continue with the usual regimen of administration of all medications related to Ovarian Stimulation
  Interventions: Drug: Ganirelix

INTERVENTIONS:
Drug: Ganirelix — Ganirelix is a GnRH antagonist, which modulates the hypothalamic-pituitary-gonadal axis by competitively binding to GnRH receptors in the pituitary gland. Consequently, there is a reversible, intense, and rapid suppression of endogenous gonadotropin release. Ganirelix is indicated for the prevention of premature luteinizing hormone (LH) surges in women undergoing controlled ovarian hyperstimulation (COH) for assisted reproductive techniques (ART).
  Arms: GnRH antagonists - control group
Drug: Medroxyprogesterone Acetate 10 MG — Medroxyprogesterone acetate is a synthetic progestin (structurally related to progesterone) with antiestrogenic, antiandrogenic, and antigonadotropic action. It inhibits pituitary gonadotropins (FSH and LH) with consequent inhibition of follicular maturation and ovulation . Medroxyprogesterone acetate is active orally and parenterally, 15 times more potent than progesterone. In addition to inhibiting ovulation, progestins also act on the endometrium preventing implantation and increasing the viscosity of cervical mucus, which hinders sperm progression in the uterus. It also transforms a proliferative endometrium into a secretory endometrium, provided that the woman has adequate endogenous estrogen levels.
  Arms: PPOS - study group

SUMMARY:
The PPOS protocol (Progestin-primed Ovarian Stimulation) involves avoiding ovulation during ovarian stimulation with progesterone. It is a reliable and safe protocol that has been widely used in recent years for in vitro fertilization, as it reduces the number of injections needed during controlled ovarian stimulation and is more cost-effective for patients.

The aim of this study is to compare two methods of ovarian stimulation for in vitro fertilization: the PPOS protocol (Group A) and the conventional protocol with injected antagonists (Group B). The goal is to determine whether both methods are equally effective in obtaining euploid embryos in the context of double ovarian stimulation.

DETAILED DESCRIPTION:
Hypothesis:

Hypothesis: The number of euploid embryos obtained in a DUOSTIM cycle with PPOS is not inferior to that obtained with the use of antagonists.

General and Specific Objectives

Main Objective: To study if there is a difference in the number of euploid embryos obtained in two groups of patients undergoing embryo accumulation for PGT-A through double ovarian stimulation, comparing two methods of pituitary suppression: Progesterone use from the start of stimulation and the use of GnRH antagonists.

Secondary Objectives:

Evaluate if there are differences between both groups regarding the number of MII oocytes.

Evaluate if there are differences between both groups regarding the number of cumulus-oocyte complexes (COC).

Study the differences between both groups regarding the total consumption of gonadotropins.

Evaluate if there are differences between both groups regarding the number of stimulation days.

Evaluate if there are differences in fertilization rate after microinjection. Evaluate if there are differences between both groups regarding the cancellation rate.

Evaluate if there are differences between both groups regarding the number of total embryos.

Evaluate if there are differences between both groups regarding the number of embryos subjected to trophectoderm biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Regular menstrual cycles between 21 and 35 days, inclusive.
* Indication of IVF with PGT-A.
* Both ovaries present.
* Ability to participate and complete the study.
* Give and sign the consent to participate in the study.

Exclusion Criteria:

* Endometriosis grade III/IV
* Concurrent participation in another study

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Euploid Embryos | From date of randomization until the end of the treatment. Assessed up to 12 weeks.
  Total number of euploid embryos after the two egg retrievals

SECONDARY OUTCOMES:
Number of Oocytes retrieved | From date of randomization until the end of the treatment. Assessed up to 12 weeks.
  Total number of oocytes retrieved after the two egg retrievals
Number of Metaphase II oovcytes | From date of randomization until the end of the treatment. Assessed up to 12 weeks.
  Total number of metaphase II oocytes retrieved after the two egg retrievals
Number of Fertilized Oovytes | From date of randomization until the end of the treatment. Assessed up to 12 weeks.
  Total number of fertilized oocytes after the two egg retrievals
Number of Blastocysts | From date of randomization until the end of the treatment. Assessed up to 12 weeks.
  Total number of blastocyst stage embryos after the two egg retrievals

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Martinez F, Rodriguez-Purata J, Beatriz Rodriguez D, Clua E, Rodriguez I, Coroleu B. Desogestrel versus antagonist injections for LH suppression in oocyte donation cycles: a crossover study. Gynecol Endocrinol. 2019 Oct;35(10):878-883. doi: 10.1080/09513590.2019.1604661. Epub 2019 May 7. PMID 31062995
- [Background] Dong M, Sun L, Huang L, Wang F, Zhang X, Liu F. Fixed Gonadotropin-Releasing Hormone Antagonist Protocol Versus Flexible Progestin-Primed Ovarian Stimulation Protocol in Patients With Asynchronous Follicular Development During Controlled Ovulation Stimulation: A Retrospective Study. Front Endocrinol (Lausanne). 2021 Nov 18;12:690575. doi: 10.3389/fendo.2021.690575. eCollection 2021. PMID 34867773
- [Background] Xiao ZN, Peng JL, Yang J, Xu WM. Flexible GnRH Antagonist Protocol versus Progestin-primed Ovarian Stimulation (PPOS) Protocol in Patients with Polycystic Ovary Syndrome: Comparison of Clinical Outcomes and Ovarian Response. Curr Med Sci. 2019 Jun;39(3):431-436. doi: 10.1007/s11596-019-2055-x. Epub 2019 Jun 17. PMID 31209815
- [Background] Giles J, Alama P, Gamiz P, Vidal C, Badia P, Pellicer A, Bosch E. Medroxyprogesterone acetate is a useful alternative to a gonadotropin-releasing hormone antagonist in oocyte donation: a randomized, controlled trial. Fertil Steril. 2021 Aug;116(2):404-412. doi: 10.1016/j.fertnstert.2021.02.036. Epub 2021 Apr 2. PMID 33814126
- [Background] Begueria R, Garcia D, Vassena R, Rodriguez A. Medroxyprogesterone acetate versus ganirelix in oocyte donation: a randomized controlled trial. Hum Reprod. 2019 May 1;34(5):872-880. doi: 10.1093/humrep/dez034. PMID 30927417
- [Background] Wang N, Zhu Q, Ma M, Liang Z, Tao Y, Wang Y, Kuang Y. Comparison of a progestin-primed ovarian stimulation protocol with a flexible GnRH antagonist protocol in patients with polycystic ovary syndrome who are participating in an IVF programme: study protocol for a randomised controlled trial. BMJ Open. 2020 Dec 2;10(12):e038153. doi: 10.1136/bmjopen-2020-038153. PMID 33268401